CLINICAL TRIAL: NCT05503992
Title: Evaluating the Efficacy of Using a Digital Consumption Tracking and Workflow Management Tool to Decrease Unmet Demand and Foster Contraceptive Continuous Use at Last Mile Point of Care in Zambia
Brief Title: Evaluating the Efficacy of Using a Digital Consumption Management Tool for Family Planning in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Pharmaceutical Systems Africa (PSA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-43082; MTaPS-19-001 (Other Grant/Funding Number: USAID)
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Family Planning
Keywords: Digital consumption management tool; Community health workers; OpenSRP; Rural Zambia

STUDY DESIGN:
Intervention Model Description: The study design is a two-arm cluster-randomized trial. The unit of randomization is the health facility catchment areas (HFCAs) which will be matched in pairs on 1) ruralness as defined by distance/time to the nearest tertiary clinic or district capital; 2) supply chain performance as defined by number of family planning commodities stockouts in the nearest preceding three to six month period for which data are available (for baseline: August to October, 2022; for endline: February to June 2023); 3) catchment area size and; 4) number of CHW affiliates. This effectiveness evaluation will be paired with a concurrent implementation evaluation, making it a Type 2 Hybrid Design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): CHWs affiliated with intervention facilities randomized to the intervention arm will be given the intervention package.
  Interventions: Other: Intervention package
- Control arm (No Intervention): CHWs affiliated with control sites randomized to the control arm will continue to implement the current standard of care which includes using paper records for inventory management and dispensing.

INTERVENTIONS:
Other: Intervention package — The intervention package will include a mobile device configured with OpenSRP configured to facilitate clinical/service provision and stock management. The intervention also incorporates a training component on OpenSRP with accompanying follow-up supervisory visits for a limited period. Per the theory of changes, these activities will improve CHWs' knowledge and ability to use the platform for clinical care, dispensing, and workflow management, leading to an improved stock of commodities to meet preferred FP needs among last mile women.
  Arms: Intervention arm

SUMMARY:
The primary objective of this evaluation is to understand the effectiveness of the OpenSRP platform on unmet family planning (FP) demand in rural Zambia. The specific objectives are to:

1. assess the impact of the intervention on satisfaction and use of modern family planning methods among last-mile people of childbearing potential; and
2. understand the impact of the intervention on FP inventory management and dispensing.

The investigators will employ mixed-methods for data collection for this two-arm cluster-randomized trial. This effectiveness evaluation will be paired with a concurrent implementation evaluation, making it a Type 2 Hybrid Design.

For the impact evaluation data will be collected from two main sources at both baseline and endline: 1) existing stock management records (eLMIS and paper records, depending on study arm); and 2) Short phone surveys with people of childbearing potential in the community.

DETAILED DESCRIPTION:
Rural health facilities catchment areas (HFCAs) and their affiliated CHWs (clusters) will be randomly assigned to the intervention or control arm. The impact evaluation will consist of a cross-sectional baseline assessment of a sample of women living in the catchment areas of both the intervention and control clusters. This will be followed by a six months of implementation phase (mobile device distribution to CHW, CHW training, CHW utilization of the Open SRP). At endline after six months, a new cross-sectional sample of respondents will be assessed in both the intervention and control clusters.

To achieve objective 1, a short questionnaire will be administered over the phone to a cross-sectional sample of last-mile people of childbearing potential living in both the intervention and control clusters. The sample will be drawn from the CHW's client lists and use a short telephone call to reach respondents.

To achieve objective 2, the same quantitative indicators will be abstracted from two different data sources, depending on the study arm: 1) OpenSRP data captured in the CHW tablets among the intervention sites, and 2) data extracted from the paper records maintained by the CHWs or the health facility or the electronic management system in the control sites (and at baseline).

ELIGIBILITY:
Inclusion Criteria:

* Resident in a study health facility catchment area (HFCA)
* Family planning (FP) client of community health worker (CHW) affiliated with one of the study sites
* Access to a mobile phone

Exclusion Criteria:

* Unwilling or unable to consent
* Currently pregnant
* Currently breastfeeding

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2523 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Percentage of women using preferred family planning method | 6 months
  Percentage of women who are still using a FP method they had obtained through the CHW or as result of referral by the CHW at the index visit.

SECONDARY OUTCOMES:
Resupply of family planning of choice | 6 months
  Percentage women whose method required re-supply were re-supplied, or received a referral for information and services specific to their method of choice, during the follow-up or secondary visit

OTHER OUTCOMES:
Stock of family planning available at health facility | 6 months
  Percentage of family planning products that are stocked out at the health facility

CONTACTS AND LOCATIONS:
Overall Officials: Veronika J Wirtz, BPharm, PhD, Principal Investigator — Boston University School of Public Health, Global Health
Locations (3):
- Zambia (3):
  - Kawambwa District Health Office, Kawambwa
  - Mansa District Health Office, Mansa
  - Samfya District Health Office, Samfya

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT05503992/ICF_000.pdf